CLINICAL TRIAL: NCT03593122
Title: Multicentric Study on the Application of WO 2085 Moisturising Cream for Breast Cancer Patients Suffering From the Symptoms of Vulvovaginal Dryness
Brief Title: Investigation on the Efficacy of WO 2085 Moisturising Cream for Breast Cancer Patients Suffering From Vulvovaginal Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: Dr. Dimitrios Chatsiproios (Unknown); Dr. med. Klaus König (Unknown); SAM®, Statistische Analysen und Monitoring GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VFAU-13/2009
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vulvovaginal Dryness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WO 2085 Moisturising Cream (Experimental): WO2085 is a hormone-free Moisturizing Cream and is used to treat "vulvovaginal dryness" symptoms.
  Interventions: Device: WO2085 Moisturising Cream

INTERVENTIONS:
Device: WO2085 Moisturising Cream — Week 1: 2.5 g of the investigational product WO2085 Moisturising Cream will be applied intravaginally, once daily in the evening. In addition 0.5 g (1 fingertip unit) may be applied to the outer genital area as needed (also several times per day).
  Week 2-4: The frequency may be reduced by the patient as needed. In addition 0.5 g (1 fingertip unit) may be applied to the outer genital area as needed (also several times per day).

SUMMARY:
The aim of the study is to gain further experience with regard to the performance of the medical device WO2085 Moisturising Cream for breast cancer patients undergoing chemotherapy or treatment with anti-oestrogens / aromatase inhibitors

DETAILED DESCRIPTION:
The goal of this application study was to answer the question as to whether the application of WO2085 Moisturising Cream for breast cancer patients undergoing chemotherapy or treatment with anti-oestrogens / aromatase inhibitors can result in an improvement in the subjective symptoms and objective diagnoses of vulvovaginal dryness while also ensuring good tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer undergoing chemotherapy OR therapy with aromatase inhibitors or anti-oestrogens (either at present or up to 3 months after ending treatment) AND with symptoms of vulvovaginal dryness since the start of tumour treatment
* Written declaration of consent for the voluntary participation in the study is present

Exclusion Criteria:

* Women who suffered symptoms of vulvovaginal dryness prior to the start of tumour treatment
* Patients undergoing radiation therapy
* Patients with other tumours
* A current vaginal infection
* Medical conditions related to the vulva or vagina
* Current additional therapy of vulvovaginal dryness or vulvovaginal atrophy
* Women who are not able to participate properly in this study
* Current alcohol and/or drug abuse
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-01-04 (Actual); Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of subjective vulvovaginal atrophy symptoms (e.g. feeling of dryness, itching) | Baseline, after 4 weeks
  Each symptom is rated according to severity on a scale from 0 to 4 (0=not present, 1=hardly pronounced, 2=moderately pronounced, 3=quite pronounced, 4=very pronounced)

SECONDARY OUTCOMES:
Change from Baseline of objective vulvovaginal atrophy symptoms (e.g. thinning of the vaginal epithelium, redness) | 4 weeks
  Each symptom is rated according to severity on a scale from 0 to 4 (0=not present, 1=hardly pronounced, 2=moderately pronounced, 3=quite pronounced, 4=very pronounced)
Global judgement of efficacy | 4 weeks
  The global judgement of efficacy will be assessed by the investigator and the patient according to the following scale: 1=very good to 6=unsatisfactory.
Global judgement of tolerability | 4 weeks
  The global judgement of tolerability will be assessed by the investigator and the patient according to the following scale: 1=very good to 6=unsatisfactory.
Adverse Events | after 4 weeks
  Adverse events will be documented on Visit after 4 weeks (and in the patient diary, if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Christoph Abels, MD, PhD, Study Director — Dr. August Wolff GmbH & Co. KG Arzneimittel
Locations (17):
- Germany (17):
  - Axel Gerick, Aachen
  - Sibylle Kaßpohl, Alzenau in Unterfranken
  - Jörg Schilling, Berlin
  - Axel Widing, Berlin
  - Alexandra Coumbos, Berlin
  - Amin Mortazawi, Darmstadt
  - Kathrin von Ardenne, Dresden
  - Joachim Larbig, Fulda
  - Nidal Gazawi, Leipzig
  - Elke Wierick, Lohsa
  - Dagmar Guth, Plauen
  - Wolfgang Clemens, Stolberg
  - Carsten Hielscher, Stralsund
  - Christopher Wolf, Ulm
  - Heidi Massinger-Biebl, Waldkirchen
  - Klaus Doubek, Wiesbaden
  - Anja Obermeyer, Würselen